CLINICAL TRIAL: NCT03759093
Title: Phenotypic Personalized Medicine: Systematically Optimized Combination Therapy in Multiple Myeloma Using CURATE.AI
Brief Title: CURATE.AI Optimized Modulation for Multiple Myeloma
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National University Hospital, Singapore (Other)
Collaborators: National University of Singapore (Other)
Responsible Party: Principal Investigator, Haematology-Oncology, Professor Chng Wee Joo, National University Hospital, Singapore
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2015/00280
Record Dates: First submitted 2018-11-20; First posted 2018-11-29 (Actual); Last update posted 2023-09-06 (Actual); Status verified 2023-08

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Bortezomib; Cyclophosphamide; Dexamethasone; Thalidomide; Lenalidomide

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard of Care (Active Comparator): Dosing of VCD(bortezomib, cyclophosphamide,dexamethasone), VTD (bortezomib,thalidomide, dexamethasone), or VRD (Bortezomib, Lenalidomide, Dexamethasone) combinations according to standard of care
  Interventions: Drug: Bortezomib; Drug: Cyclophosphamide; Drug: Dexamethasone; Drug: Thalidomide; Drug: Lenalidomide
- CURATE.AI-guided dosing (Experimental): CURATE.AI optimized modulation of bortezomib and cyclophosphamide dosages in the VCD (bortezomib, cyclophosphamide, dexamethasone), bortezomib and thalidomide in the VTD (bortezomib, thalidomide, dexamethasone) or bortezomib and lenalidomide in the VRD (bortezomib, lenalidomide, dexamethasone) combinations
  Interventions: Other: CURATE.AI-Guided dosage modulation; Drug: Bortezomib; Drug: Cyclophosphamide; Drug: Thalidomide; Drug: Dexamethasone; Drug: Lenalidomide

INTERVENTIONS:
Drug: Bortezomib — Standard dosing based on product insert and subjected to dose adjustments as determined by clinical care team
  Other Names: Velcade
  Arms: Standard of Care
Drug: Cyclophosphamide — Standard dosing based on product insert and subjected to dose adjustments as determined by clinical care team
  Arms: Standard of Care
Drug: Dexamethasone — Standard dosing based on product insert and subjected to dose adjustments as determined by clinical care team
  Arms: Standard of Care
Other: CURATE.AI-Guided dosage modulation — CURATE.AI-guided modulation of Velcade and Cyclophosphamide dosages for VCD regimen, Velcade and Thalidomide dosages for VTD regimen, and Velcade and Lenalidomide dosages for VRD regimen
  Arms: CURATE.AI-guided dosing
Drug: Thalidomide — Standard dosing based on product insert and subjected to dose adjustments as determined by clinical care team
  Arms: Standard of Care
Drug: Bortezomib — Dose in a range of 0.7,1.0,1.3 mg/m2 subcutaneous (SC) injection on Day 1, 8, 15 ,22 for cycles 1 to 4 , as determined and guided by CURATE.AI and approved by the clinical care team
  Other Names: Velcade
  Arms: CURATE.AI-guided dosing
Drug: Cyclophosphamide — Dosing in a range of 100, 300, 500 mg PO on Day 1, 8, 15, 22 for cycles 1 to 4 as determined and guided by CURATE.AI and approved by the clinical care team.
  Arms: CURATE.AI-guided dosing
Drug: Thalidomide — Dose in a range of 50-200mg PO on day 1-28 for cycles 1 to 4 as determined and guided by CURATE.AI and approved by the clinical care team.
  Arms: CURATE.AI-guided dosing
Drug: Dexamethasone — 40 mg PO on Day 1 ,8 , 15, 22 for cycles 1 to 4, as determined and guided by the clinical care team according to standard of care
  Arms: CURATE.AI-guided dosing
Drug: Lenalidomide — Standard dosing based on product insert and subjected to dose adjustments as determined by clinical care team
  Other Names: Revlimid
  Arms: Standard of Care
Drug: Lenalidomide — Dose in a range of 5-25mg PO on day 1-21 for cycles 1 to 4, as determined and guided by CURATE.AI and approved by the clinical care team.
  Other Names: Revlimid
  Arms: CURATE.AI-guided dosing

SUMMARY:
Clinical trial applying CURATE.AI, a Phenotypic Precision Medicine (PPM) platform, to Bortezomib, Thalidomide, Cyclophosphamide and Lenalidomide dosing in multiple myeloma patients to show improvement in response.

DETAILED DESCRIPTION:
In conventional combination chemotherapy, drug doses are typically determined using dose escalation to reach a maximum tolerated dose (MTD) or via dose expansion to identify suitable regimen administration guideline, and the combinations are subsequently administered at fixed doses. During the course of treatment, the patient's response to therapy evolves and changes due to the time-dependent, dose dependent, and patient-specific nature of drug synergy and resulting efficacy and tolerability. To overcome this challenge, we have developed CURATE.AI, a Phenotypic Precision Medicine (PPM) platform, which has been clinically validated and used to prospectively optimize patient liver transplant immunosuppression, and tuberculosis therapy, among other indications. In this study, CURATE.AI may improve patient response by providing dose recommendations for Bortezomib, Thalidomide, Cyclophosphamide and Lenalidomide to the clinical team over the course of the patient's treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Multiple myeloma diagnosed according to standard criteria, without prior anti-myeloma treatment at study entry. Both transplant eligible and ineligible patients may be included.
2. Patients must have evaluable multiple myeloma with at least one of the following (within 21 days of starting treatment)

   1. Serum M-protein ≥ 0.5g/dL, or
   2. In subjects without detectable serum M-protein, Urine M-protein ≥ 200mg/24 hour, or serum free light chai (sFLC) > 100mg/L (involved light chain) and an abnormal kappa/Lambda ratio
3. Males and females ≥ 18 years of age or > country's legal age for adult consent
4. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 to 2
5. Patients must meet the following clinical laboratory criteria with 21 days of starting treatment:

   1. Absolute neutrophil count (ANC) ≥ 1,000/mm3 and platelet ≥ 50,000/mm3 (≥ 30,000/mm3 if myeloma involvement in the bone marrow is >50%)
   2. Total bilirubin ≤ 1.5 x the upper limit of the normal range (ULN). Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 3 x ULN.
   3. Calculated creatinine clearance ≥ 30mL/min or creatinine < 3mg/dL.
6. Written informed consent in accordance with federal, local and institutional guidelines

Exclusion Criteria:

1. Female patients who are lactating or pregnant
2. Multiple Myeloma of IgM subtype
3. Glucocorticoid therapy (prednisolone > 30mg/day or equivalent) within 14 days prior to informed consent obtained
4. POEMS syndrome
5. Plasma cell leukaemia or circulating plasma cells ≥ 2 x 109/L
6. Waldenstrom's Macroglobulinaemia
7. Patients with known amyloidosis
8. Chemotherapy with approved or investigation anticancer therapeutics within 21 days prior to starting bortezomib treatment
9. Focal radiation therapy within 7 days prior to start of treatment. Radiation therapy to an extended field involving a significant volume of bone marrow within 21 days prior to start of treatment
10. Immunotherapy (excluding steroids) 21 days prior to start of treatment
11. Major surgery (excluding kyphoplasty) within 28 days prior to start of treatment
12. Active congestive heart failure (New York Heart Association [NYHA] Class III or IV), symptomatic ischaemia, or conduction abnormalities uncontrolled by conventional intervention. Myocardial infarction within 4 months prior to informed consent obtained
13. Known HIV seropositive, hepatitis C infection, and/or hepatitis B (except for patients with hepatitis B surface antigen or core antibody receiving and responding to antiviral therapy directed at hepatitis B: these patients are allowed)
14. Patients with known cirrhosis
15. Second malignancy within the past 3 years except:

    1. Adequately treated basal cell or squamous cell skin cancer
    2. Carcinoma in situ of the cervix
    3. Breast carcinoma in situ with full surgical resection
16. Patients with myelodysplastic syndrome
17. Patients with steroid, cyclophosphamide, bortezomib, lenalidomide or thalidomide hypersensitivity
18. Patients with a calculated creatinine clearance less than 30ml/min by the Cockroft Galt method.
19. Prior treatment with Bortezomib
20. Contraindication to any of the required concomitant drugs or supportive treatments
21. Any clinically significant medical disease or psychiatric condition that, in the investigator's opinion, may interfere with protocol

Ages: 21 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-09-10 (Estimated); Primary Completion 2025-09-10 (Estimated); Study Completion 2025-09-10 (Estimated)

PRIMARY OUTCOMES:
Response rate | Up to 16 weeks or at the end of cycle 4 of treatment (each cycle is 28 days)
  Complete response (CR), or stringent complete response (sCR), or very good partial response (VGPR), or partial response (PR) based on IMWG criteria at the end of cycle 4

SECONDARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events (Safety and Tolerability) | Up to 16 weeks or at the end of cycle 4 of treatment (each cycle is 28 days)
  Occurrence of adverse events throughout the study, graded via Common Terminology Criteria for Adverse Events (CTCAE) v 4.03 criteria.

CONTACTS AND LOCATIONS:
Locations (1):
- National University Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pantuck, A.J., Lee, D.K., Kee, T., Wang, P., Lakhotia, S., Silverman, M.H., Mathis, C., Drakaki, A., Belldegrun, A.S., Ho, C.M. and Ho, D., 2018. Modulating BET Bromodomain Inhibitor ZEN-3694 and Enzalutamide Combination Dosing in a Metastatic Prostate Cancer Patient Using CURATE. AI, an Artificial Intelligence Platform. Advanced Therapeutics, 1(6), p.1800104.